CLINICAL TRIAL: NCT05782400
Title: Multiomics Approach for Patients Stratification and Novel Target Identification in Metastatic Clear Renal Cell Carcnoma
Brief Title: Multiomics Approach in Metastatic Clear Renal Cell Carcnoma
Status: Active, not recruiting | Type: Observational
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Principal Investigator, Giuseppe Procopio, Director of Genitourinary Medical Oncology, Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Other Study IDs: INT220-22
Record Dates: First submitted 2023-02-10; First posted 2023-03-23 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Metastatic Clear Cell Renal Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * FFPE samples will be collected at baseline and, when feasible, at the first progression of the disease (PD). FFPE specimens will be sent to the coordinator site (INT). A centralized designated expert pathology will review these specimens to confirm the diagnosis and to identify regions of interest. mRNA and DNA sequencing will be used to dissect the molecular and genomic profiles of this cohort.
  * Blood samples will be collected at baseline, at 1 month and at the first PD. Sixteen ml of blood will be collected in EDTA tubes and centrifuged at 1900×g for 10 min at 4 °C within 2 h after drawing to collect plasma, which will be stored at -80°C until analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: CT scan — CT scan at baseline and then every three months as per clinical practice. The standardization of the procedure of images' collection through a CT- acquisition's protocol has been planned to control bias.
Biological: Plasma collection — ● Blood samples will be collected at baseline, at 1 month and at the first PD. Sixteen ml of blood will be collected in EDTA tubes and centrifuged at 1900×g for 10 min at 4 °C within 2 h after drawing to collect plasma, which will be stored at -80°C until analysis. Plasma samples will be sent to the Laboratory of Pharmacogenetics - Unit of Clinical Pharmacology and Pharmacogenetics - University Hospital of Pisa. Plasma samples will be used to isolate cell free DNA (cfDNA) and microvesicles-derived RNA for molecular analysis.

SUMMARY:
The choice of the best strategy in treatment-naive metastatic clear-cell renal cell carcinoma (mccRCC) patients is becoming an issue, since no biomarkers are available to guide the treatment allocation strategy. The elucidation of predictive factors to develop tailored strategies of treatment is an urgent unmet clinical need. Recently there has been a great deal of interest in non-invasive liquid biopsy methods for their ability to detect and characterize circulating cell-free DNA (cfDNA), extracellular vescicles associated RNAs and circulating tumor cells and to allow longitudinal evaluation of tumor evolution. An additional field of intense research is also radiomics as a novel approach to develop predictive tools by correlating imaging features to tumor characteristics including histology, tumor grade, genetic patterns and molecular phenotypes, as well as clinical outcomes in patients with renal neoplasms.

The use of computational approaches to integrate informations, obtained from genomic and transcriptomic analysis of neoplastic tissues and of cfDNA) or microvescicle-associated RNA in blood and from radiomics, can be exploited to define an optimal allocation strategy for patients with mccRCC undergoing first-line therapy and to identify novel targets in mccRCC.

Aims of the study are: to identify molecular subtypes, signatures or biomarkers in mccRCC associated with different clinical outcome by applying bioinformatic analysis; to extract descriptive features in mccRCC from radiological imaging data; to integrate omics-driven and clinic-pathological characteristics with radiomic features extracted from the tumor and tumor environment to inform on biological features relevant to therapy outcome.

This multicentric prospective study will evaluate genomics and radiomics in treatment-naïve advanced ccRCC patients. 100 eligible patients will be identified after screening, candidate to receive first-line treatment as investigator choice per clinical practice. Tissue and plasma samples and CT exams will be collected at different intervals to provide a comprehensive molecular profile and radiomic features extrapolation, respectively. Artificial neural networks will be used to build a genomic-radiomic profile of patients to correlate to treatment response. This sample size will allow an exploratory analysis of the prognostic and predictive performance of the multiomic classifier, to be subsequently validated in a larger expansion cohort of patients.

DETAILED DESCRIPTION:
IMPACT In the last ten years the systemic treatment of metastatic renal cell carcinoma has been revolutioned with the introduction of at least ten active drugs. With the advent of novel immuno-based and tyrosine kinase inhibitors (TKIs)-based combinations, the choice of the best strategy in treatment-naive metastatic clear-cell renal cell carcinoma (mccRCC) patients (pts) is becoming an issue, since no biomarkers are available to guide the treatment allocation strategy . In recent clinical trials, combination therapies including nivolumab plus ipilimumab, pembrolizumab plus axitinib, atezolizumab plus bevacizumab, avelumab plus axitinib, pembrolizumab plus lenvatinib and nivolumab plus cabozantinib exhibited significant benefits in terms of overall survival (OS) and/or progression-free survival (PFS) for mRCC compared with sunitinib as a standard first-line treatment for mRCC . However, there is a clear need for clinical predictive biomarkers to guide optimal treatment decisions. Through the above research the investigators are confident to provide proof of concept that combine the informations from genomics and radiomics using computational approaches such as machine learning, will provide an opportunity for a molecularly driven patient's stratification.

RATIONALE AND FEASIBILITY

BIOMARKERS Risk stratification models based on gene expression pattern (both messenger and long non-coding RNA) in ccRCC have proven to have strong prognostic values. Hence, there is an interest in the identification and development of treatment predictive biomarkers to enable precision oncology increasing drug response. Multiple candidates for predictive biomarkers from plasma, tumor, and host tissues have been explored in patients with metastatic renal-cell carcinoma who are receiving systemic therapies, but, as yet, none have entered clinical practice and all require prospective validation in clinical trials.

In the era of VEGF inhibitors, the investigators counted on IMDC (International Metastatic RCC Database Consortium) model, considering Karnofsky performance status <80, time to initiation of therapy <1 year, hemoglobin < lower level of normal, serum calcium, neutrophil count, and platelet count > upper limit of normal. CheckMate 214 study showed that OS and ORR were significantly higher with nivolumab plus ipilimumab than with sunitinib among intermediate- and poor-risk pts. Extended study follow-up of KEYNOTE-426 study demonstrated that the benefit in OS and PFS is consistent in this class of patients's risk also with the IO/TKI combination therapy. The IMDC score is confirmed to be prognostic in every combos study.

PD-L1 has also been demonstrated to be a prognostic marker for poor prognosis in RCC, regardless of the type of treatment used. More recently PD-L1 expression has also been evaluated for its predictive role that is only partially confirmed in the CheckMate-214 population that received IO-IO combo and considered a poor marker for targeted therapies. Gene signatures from ImMotion 150 and 151 evidenced that two different signatures (angiogenesis versus immune signature) in RCC patients could predict the response to combo treatment.

Metabolomics have also been assessed as potential biomarkers for RCC giving new insights into the understanding of RCC clinical behavior and for the development of new therapeutic strategies. Both tumor tissue and blood are interesting source for the study of potential biomarkers. Plasma samples in particular have been analyzed to better understand the role of components of the proangiogenic and cellular proliferation pathways. Another topic is the study of cytokines, circulating endothelial cells, and gene expression controlling mechanisms. Moreover, germline genetic variations in important genes related to drug mechanism-of-action and metabolism have been under investigation as well as factors implicated in gene expression regulation by epigenetic mechanisms or by post-transcriptional regulation.

RADIOMICS Computed tomography (CT) is widely available, routinely used in the care of patients with metastatic tumors treated with antiangiogenic therapy and yields quantitative digital data. Many studies have used CT noninvasive imaging-based methods to assess the pathologic grade of renal tumor before surgery. Various radiological features such as tumor size and pattern enhancement have been shown to correlate with tumor grade. However, it is difficult to predict the pathologic grade of renal tumor with only information obtained from traditional radiologic features. Conversely, radiomics analysis involves the automatic extraction of data not recognizable to the human eye resulting in highly detailed imaging features regarding tumor structure, shape and image intensity. Radiomics may provide a novel approach to develop predictive tools by correlating imaging features to tumor characteristics including histology, tumor grade, genetic patterns and molecular phenotypes, as well as clinical outcomes. Extracting data from imaging the aim is to provide information beyond what can be achieved from human imaging interpretation alone.

In clinical practice, the prediction of RCC aggressiveness through imaging findings remains a challenge. A retrospective study by Shu et al. demonstrated that radiomics features could be used as biomarkers for the preoperative evaluation of the ccRCC Fuhrman grades. In the post-treatment setting, radiomics may assist in predicting a response to systemic therapy, including to antiangiogenic treatment, which may not be adequately assessed with traditional size-based criteria.

Smith and colleagues used a custom post-processing software and algorithm to develop a novel system to quantify changes in the amount of vascularized tumor within specific attenuation thresholds, termed the vascular tumor burden. This semi automated biomarker, in addition to other tumor metrics, such as length, area, and mean attenuation, were used to predict response to antiangiogenic therapy with sunitinib. Changes in the vascular tumor burden metric on initial post-therapy imaging after the initiation of sunitinib showed a better separation of progression free survival between non-responders and responders compared with other commonly used response criteria changes in tumor metrics, including length, area, mean attenuation, RECIST, CHOI, modified CHOI, MASS, and 10% sum long diameter. Extension of radiomic analysis through radiogenomics, radiometabolomics, and correlation with other epidemiologic, clinical, and tissue-based datasets have the potential to improve patient management in the era of personalized medicine. Understanding what these technologies can offer will allow radiologists to play a larger role in the care of patients with RCC.

CT dynamic contrast-enhanced is a capable tool to quantify tumor enhancement and its response to anti-angiogenetic therapies. Han et al found a correlation between tumor renal enhancement at baseline and response and PFS after treatment with sunitinib or sorafenib. In contrast, other studies have demonstrated that although the perfusion parameters at baseline were higher in patients with longer survival times, they were not significantly predictive of outcome, except when a cut-off analysis was established. Other CT-based methods for assessing tumor response to anti-angiogenic therapy and predicting clinical outcome are undergoing further evaluation. Among them, radiomics CT features such as heterogeneity, entropy, and texture uniformity are additional parameters that show promise for assessing the anti-angiogenic response of metastatic renal cell carcinoma. The correlation of these imaging data with genomics (ie, radiogenomics), metabolomics (ie, radiometabolomics) and beyond, offers an opportunity to generate objective, quantitative biomarkers of tumor biology that may be used to predict patient's prognosis and likelihood of response to therapy, overcoming some of the challenges associated with disease heterogeneity.

ARTIFICIAL INTELLIGENCE Artificial intelligence systems, in particular those based on Machine Learning and Deep Learning, are able to autonomously identify salient patterns and complex relationships among data by just looking at sample populations. Their ability to process heterogeneous data, for both classification and prediction purposes, may provide a valid contribution to better stratify RCC patients. Recently, some works have attempted to use Machine and Deep Learning for the differentiation between benign and malignant small renal masses, based on textural analysis of CT scans, for the prediction of the Fuhrman nuclear grade, and gene expression-based molecular signatures.

Overall, the stratification of RCC patients still remains a challenging task, especially when considering the molecular heterogeneity of kidney tumors.

The ability to combine the information from genomics and radiomics using computational approaches based on Machine Learning, provides an opportunity to re-classify patients into subgroups that could better guide treatment strategies. Both supervised and unsupervised techniques can be used to identify a biomarker signature-score as well as to predict response/resistance to therapies.

PRELIMINARY DATA The investigators have preliminary biological data on blood samples of 32 mRCC patients obtained at treatment baseline. The majority of patients received as first line the combination of nivolumab and ipilimumab, 9 patients received sunitinib, 5 were administered with pazopanib, and 6 patients received cabozantinib. The molecular analysis was conducted using the NGS OncoMine Solid Tumor Panel (Thermo Fisher). Twentyfive patients (78,1%) were carriers of a molecular alteration in one or more genes including: TP53, mTOR, PIK3CA, BRAF, EGFR, RET, GNAS, SF3B1, PDGFRA. The reported allele frequency ranged between 3% and 12%. The preliminary analysis shows that patients with multiple mutations have a better response (PR+SD vs PD) from immunotherapy.

EXPERIMENTAL DESIGN This is a multicentric prospective translational study evaluating genomics and radiomics in treatment- naïve advanced ccRCC pts candidate to receive first-line systemic therapy. Nine centers in Italy, including: Istituto Nazionale dei Tumori (INT) of Milan, European Institute of Oncology (IEO) of Milan, Istituto Oncologico Veneto (IOV), Policlinico San Martino of Genova, Istituto Nazionale dei Tumori of Napoli, University Hospital of Parma, Humanitas Research Hospital of Milan, Oncological Center of Aviano and Fondazione Policlinico Universitario Agostino Gemelli of Rome will be involved in the accrual and the treatment of patients.

ELIGIBILITY:
INCLUSION CRITERIA:

* Signed Written Informed Consent
* Male or female subjects aged ≥18 years old
* Histologically confirmed advanced/metastatic RCC with predominantly clear-cell subtype
* Previous nephrectomy is permitted
* Availability of tumor tissue sample for biomarker analysis
* Advanced (not amenable to curative surgery or radiation therapy) or metastatic (AJCC Stage IV) RCC, candidate to receive first-line systemic treatment with monotherapy TKI or IO+TKI or IO+IO
* No prior systemic therapy for RCC with the following exception: prior adjuvant therapy for completely resectable RCC (concluded at least 6 months before study entry)
* All IMDC risk (good, intermediate, poor)
* TC scan performed with and without contrast medium, at baseline (according to protocol guidelines as reported below in Table 1)
* At least one measurable lesion as defined by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
* Eastern Cooperative Oncology Group performance status 0 or 1
* Capable of understanding and complying with the protocol requirements.

EXCLUSION CRITERIA:

* Any prior systemic treatment for RCC in the advanced/metastatic settings
* Prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways
* Previous exposure to tyrosine kinase inhibitors in the advanced/metastatic settings
* Active seizure disorder or evidence of brain metastases, spinal cord compression, or carcinomatous meningitis
* Diagnosis of any non-RCC malignancy occurring within 2 years prior to the date of the start of treatment except for adequately treated basal cell or squamous cell skin cancer, or carcinoma in situ of the breast or of the cervix or low-grade prostate cancer (≤pT2, N0; Gleason 6) with no plans for treatment intervention
* Radiation therapy for bone metastasis within 2 weeks, any other external radiation therapy within 4 weeks before the start of treatment. Subjects with clinically relevant ongoing complications from prior radiation therapy are not eligible.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients (nr 100) diagnosed with advanced RCC with predominantly clear-cell subtype, candidate to receive first-line systemic treatment as per clinical practice (investigators choice).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-02-28 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Blood and tissue analysis | 36 Months
  Investigation of the predictive role of circulating miRNAs and gene alterations in patients who respond to first-line treatments versus those who do not respond before treatment, after 1 month (4 weeks), after 3 months (12 weeks), and at the time of disease progression. Tissue and blood samples will be studied with Illumina NextSeq 500 platform and analyzed with the GeneGlobe online software. Methods that combine different clustering algorithms and gene variability metrics will be used to identify robust mccRCC molecular subtypes from expression data and to investigate their association with clinical outcomes.

SECONDARY OUTCOMES:
Radiomics analysis | 36 Months
  Characterization of alterations in radiological imaging data in mRCC in radiological imaging data in mRCC through CT segmentation. Through open-source software analysis, we aim to extrapolate from the image patterns of quantitative characteristics (features) not visible to the naked eye, compare different images of the same disease with known diagnosis (ground truth), and develop a predictive computational model of disease. CT scan for Radiomics will be performed at baseline and every three months.

OTHER OUTCOMES:
Computational analysis of mutational, transcriptomic and radiomic data | 48 Months
  Radio-genomic analysis to identify a Radiomics and a molecular score. An artificial neural network-based approach to creating a combined Genomic plus Radiomics signature. Integration of high-dimensional data obtained with clinical data. For this task, we will incorporate NGS and Radiomics datasets to develop an ad hoc AI-based classification model able to efficiently merge and evaluate the array of available information. The achieved biotechnological signature of mccRCC and its evolution over time will also be assessed to suggest an easily interpretable predictive tool (nomogram) of clinical outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Procopio, MD, Principal Investigator — Fondazione IRCCS istituto Nazionale dei Tumori di Milano
Locations (1):
- Istituto Tumori, Milan, Mi, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Choueiri TK, Motzer RJ. Systemic Therapy for Metastatic Renal-Cell Carcinoma. N Engl J Med. 2017 Jan 26;376(4):354-366. doi: 10.1056/NEJMra1601333. No abstract available. PMID 28121507
- [Background] Motzer RJ, Tannir NM, McDermott DF, Aren Frontera O, Melichar B, Choueiri TK, Plimack ER, Barthelemy P, Porta C, George S, Powles T, Donskov F, Neiman V, Kollmannsberger CK, Salman P, Gurney H, Hawkins R, Ravaud A, Grimm MO, Bracarda S, Barrios CH, Tomita Y, Castellano D, Rini BI, Chen AC, Mekan S, McHenry MB, Wind-Rotolo M, Doan J, Sharma P, Hammers HJ, Escudier B; CheckMate 214 Investigators. Nivolumab plus Ipilimumab versus Sunitinib in Advanced Renal-Cell Carcinoma. N Engl J Med. 2018 Apr 5;378(14):1277-1290. doi: 10.1056/NEJMoa1712126. Epub 2018 Mar 21. PMID 29562145
- [Background] Rini BI, Powles T, Atkins MB, Escudier B, McDermott DF, Suarez C, Bracarda S, Stadler WM, Donskov F, Lee JL, Hawkins R, Ravaud A, Alekseev B, Staehler M, Uemura M, De Giorgi U, Mellado B, Porta C, Melichar B, Gurney H, Bedke J, Choueiri TK, Parnis F, Khaznadar T, Thobhani A, Li S, Piault-Louis E, Frantz G, Huseni M, Schiff C, Green MC, Motzer RJ; IMmotion151 Study Group. Atezolizumab plus bevacizumab versus sunitinib in patients with previously untreated metastatic renal cell carcinoma (IMmotion151): a multicentre, open-label, phase 3, randomised controlled trial. Lancet. 2019 Jun 15;393(10189):2404-2415. doi: 10.1016/S0140-6736(19)30723-8. Epub 2019 May 9. PMID 31079938
- [Background] Rini BI, Plimack ER, Stus V, Gafanov R, Hawkins R, Nosov D, Pouliot F, Alekseev B, Soulieres D, Melichar B, Vynnychenko I, Kryzhanivska A, Bondarenko I, Azevedo SJ, Borchiellini D, Szczylik C, Markus M, McDermott RS, Bedke J, Tartas S, Chang YH, Tamada S, Shou Q, Perini RF, Chen M, Atkins MB, Powles T; KEYNOTE-426 Investigators. Pembrolizumab plus Axitinib versus Sunitinib for Advanced Renal-Cell Carcinoma. N Engl J Med. 2019 Mar 21;380(12):1116-1127. doi: 10.1056/NEJMoa1816714. Epub 2019 Feb 16. PMID 30779529
- [Background] Motzer RJ, Penkov K, Haanen J, Rini B, Albiges L, Campbell MT, Venugopal B, Kollmannsberger C, Negrier S, Uemura M, Lee JL, Vasiliev A, Miller WH Jr, Gurney H, Schmidinger M, Larkin J, Atkins MB, Bedke J, Alekseev B, Wang J, Mariani M, Robbins PB, Chudnovsky A, Fowst C, Hariharan S, Huang B, di Pietro A, Choueiri TK. Avelumab plus Axitinib versus Sunitinib for Advanced Renal-Cell Carcinoma. N Engl J Med. 2019 Mar 21;380(12):1103-1115. doi: 10.1056/NEJMoa1816047. Epub 2019 Feb 16. PMID 30779531
- [Background] Powles T, Plimack ER, Soulieres D, Waddell T, Stus V, Gafanov R, Nosov D, Pouliot F, Melichar B, Vynnychenko I, Azevedo SJ, Borchiellini D, McDermott RS, Bedke J, Tamada S, Yin L, Chen M, Molife LR, Atkins MB, Rini BI. Pembrolizumab plus axitinib versus sunitinib monotherapy as first-line treatment of advanced renal cell carcinoma (KEYNOTE-426): extended follow-up from a randomised, open-label, phase 3 trial. Lancet Oncol. 2020 Dec;21(12):1563-1573. doi: 10.1016/S1470-2045(20)30436-8. Epub 2020 Oct 23. PMID 33284113
- [Background] Motzer R, Alekseev B, Rha SY, Porta C, Eto M, Powles T, Grunwald V, Hutson TE, Kopyltsov E, Mendez-Vidal MJ, Kozlov V, Alyasova A, Hong SH, Kapoor A, Alonso Gordoa T, Merchan JR, Winquist E, Maroto P, Goh JC, Kim M, Gurney H, Patel V, Peer A, Procopio G, Takagi T, Melichar B, Rolland F, De Giorgi U, Wong S, Bedke J, Schmidinger M, Dutcus CE, Smith AD, Dutta L, Mody K, Perini RF, Xing D, Choueiri TK; CLEAR Trial Investigators. Lenvatinib plus Pembrolizumab or Everolimus for Advanced Renal Cell Carcinoma. N Engl J Med. 2021 Apr 8;384(14):1289-1300. doi: 10.1056/NEJMoa2035716. Epub 2021 Feb 13. PMID 33616314
- [Background] Choueiri TK, Powles T, Burotto M, Escudier B, Bourlon MT, Zurawski B, Oyervides Juarez VM, Hsieh JJ, Basso U, Shah AY, Suarez C, Hamzaj A, Goh JC, Barrios C, Richardet M, Porta C, Kowalyszyn R, Feregrino JP, Zolnierek J, Pook D, Kessler ER, Tomita Y, Mizuno R, Bedke J, Zhang J, Maurer MA, Simsek B, Ejzykowicz F, Schwab GM, Apolo AB, Motzer RJ; CheckMate 9ER Investigators. Nivolumab plus Cabozantinib versus Sunitinib for Advanced Renal-Cell Carcinoma. N Engl J Med. 2021 Mar 4;384(9):829-841. doi: 10.1056/NEJMoa2026982. PMID 33657295
- [Background] Brooks SA, Brannon AR, Parker JS, Fisher JC, Sen O, Kattan MW, Hakimi AA, Hsieh JJ, Choueiri TK, Tamboli P, Maranchie JK, Hinds P, Miller CR, Nielsen ME, Rathmell WK. ClearCode34: A prognostic risk predictor for localized clear cell renal cell carcinoma. Eur Urol. 2014 Jul;66(1):77-84. doi: 10.1016/j.eururo.2014.02.035. Epub 2014 Feb 25. PMID 24613583
- [Background] Qu L, Wang ZL, Chen Q, Li YM, He HW, Hsieh JJ, Xue S, Wu ZJ, Liu B, Tang H, Xu XF, Xu F, Wang J, Bao Y, Wang AB, Wang D, Yi XM, Zhou ZK, Shi CJ, Zhong K, Sheng ZC, Zhou YL, Jiang J, Chu XY, He J, Ge JP, Zhang ZY, Zhou WQ, Chen C, Yang JH, Sun YH, Wang LH. Prognostic Value of a Long Non-coding RNA Signature in Localized Clear Cell Renal Cell Carcinoma. Eur Urol. 2018 Dec;74(6):756-763. doi: 10.1016/j.eururo.2018.07.032. Epub 2018 Aug 22. PMID 30143382
- [Background] Havel JJ, Chowell D, Chan TA. The evolving landscape of biomarkers for checkpoint inhibitor immunotherapy. Nat Rev Cancer. 2019 Mar;19(3):133-150. doi: 10.1038/s41568-019-0116-x. PMID 30755690
- [Background] Sonpavde G, Choueiri TK. Biomarkers: the next therapeutic hurdle in metastatic renal cell carcinoma. Br J Cancer. 2012 Sep 25;107(7):1009-16. doi: 10.1038/bjc.2012.399. Epub 2012 Sep 4. PMID 22948724
- [Background] McDermott DF, Huseni MA, Atkins MB, Motzer RJ, Rini BI, Escudier B, Fong L, Joseph RW, Pal SK, Reeves JA, Sznol M, Hainsworth J, Rathmell WK, Stadler WM, Hutson T, Gore ME, Ravaud A, Bracarda S, Suarez C, Danielli R, Gruenwald V, Choueiri TK, Nickles D, Jhunjhunwala S, Piault-Louis E, Thobhani A, Qiu J, Chen DS, Hegde PS, Schiff C, Fine GD, Powles T. Clinical activity and molecular correlates of response to atezolizumab alone or in combination with bevacizumab versus sunitinib in renal cell carcinoma. Nat Med. 2018 Jun;24(6):749-757. doi: 10.1038/s41591-018-0053-3. Epub 2018 Jun 4. PMID 29867230
- [Background] Jing L, Guigonis JM, Borchiellini D, Durand M, Pourcher T, Ambrosetti D. LC-MS based metabolomic profiling for renal cell carcinoma histologic subtypes. Sci Rep. 2019 Oct 30;9(1):15635. doi: 10.1038/s41598-019-52059-y. PMID 31666664
- [Background] Lakshminarayanan H, Rutishauser D, Schraml P, Moch H, Bolck HA. Liquid Biopsies in Renal Cell Carcinoma-Recent Advances and Promising New Technologies for the Early Detection of Metastatic Disease. Front Oncol. 2020 Oct 28;10:582843. doi: 10.3389/fonc.2020.582843. eCollection 2020. PMID 33194717
- [Background] Bex A, Fournier L, Lassau N, Mulders P, Nathan P, Oyen WJ, Powles T. Assessing the response to targeted therapies in renal cell carcinoma: technical insights and practical considerations. Eur Urol. 2014 Apr;65(4):766-77. doi: 10.1016/j.eururo.2013.11.031. Epub 2013 Nov 28. PMID 24341958
- [Background] Yi X, Xiao Q, Zeng F, Yin H, Li Z, Qian C, Wang C, Lei G, Xu Q, Li C, Li M, Gong G, Zee C, Guan X, Liu L, Chen BT. Computed Tomography Radiomics for Predicting Pathological Grade of Renal Cell Carcinoma. Front Oncol. 2021 Jan 27;10:570396. doi: 10.3389/fonc.2020.570396. eCollection 2020. PMID 33585193
- [Background] Shu J, Tang Y, Cui J, Yang R, Meng X, Cai Z, Zhang J, Xu W, Wen D, Yin H. Clear cell renal cell carcinoma: CT-based radiomics features for the prediction of Fuhrman grade. Eur J Radiol. 2018 Dec;109:8-12. doi: 10.1016/j.ejrad.2018.10.005. Epub 2018 Oct 5. PMID 30527316
- [Background] Smith AD, Zhang X, Bryan J, Souza F, Roda M, Sirous R, Zhang H, Vasanji A, Griswold M. Vascular Tumor Burden as a New Quantitative CT Biomarker for Predicting Metastatic RCC Response to Antiangiogenic Therapy. Radiology. 2016 Nov;281(2):484-498. doi: 10.1148/radiol.2016160143. Epub 2016 Sep 2. PMID 27603788
- [Background] Han KS, Jung DC, Choi HJ, Jeong MS, Cho KS, Joung JY, Seo HK, Lee KH, Chung J. Pretreatment assessment of tumor enhancement on contrast-enhanced computed tomography as a potential predictor of treatment outcome in metastatic renal cell carcinoma patients receiving antiangiogenic therapy. Cancer. 2010 May 15;116(10):2332-42. doi: 10.1002/cncr.25019. PMID 20225226
- [Background] Fournier LS, Oudard S, Thiam R, Trinquart L, Banu E, Medioni J, Balvay D, Chatellier G, Frija G, Cuenod CA. Metastatic renal carcinoma: evaluation of antiangiogenic therapy with dynamic contrast-enhanced CT. Radiology. 2010 Aug;256(2):511-8. doi: 10.1148/radiol.10091362. Epub 2010 Jun 15. PMID 20551183
- [Background] Hudson JM, Bailey C, Atri M, Stanisz G, Milot L, Williams R, Kiss A, Burns PN, Bjarnason GA. The prognostic and predictive value of vascular response parameters measured by dynamic contrast-enhanced-CT, -MRI and -US in patients with metastatic renal cell carcinoma receiving sunitinib. Eur Radiol. 2018 Jun;28(6):2281-2290. doi: 10.1007/s00330-017-5220-2. Epub 2018 Jan 30. PMID 29383520
- [Background] Zhou L, Zhang Z, Chen YC, Zhao ZY, Yin XD, Jiang HB. A Deep Learning-Based Radiomics Model for Differentiating Benign and Malignant Renal Tumors. Transl Oncol. 2019 Feb;12(2):292-300. doi: 10.1016/j.tranon.2018.10.012. Epub 2018 Dec 17. PMID 30448734
- [Background] Kuusk T, Neves JB, Tran M, Bex A. Radiomics to better characterize small renal masses. World J Urol. 2021 Aug;39(8):2861-2868. doi: 10.1007/s00345-021-03602-y. Epub 2021 Jan 26. PMID 33495866
- [Background] Lin F, Cui EM, Lei Y, Luo LP. CT-based machine learning model to predict the Fuhrman nuclear grade of clear cell renal cell carcinoma. Abdom Radiol (NY). 2019 Jul;44(7):2528-2534. doi: 10.1007/s00261-019-01992-7. PMID 30919041
- [Background] Suarez-Ibarrola R, Hein S, Reis G, Gratzke C, Miernik A. Current and future applications of machine and deep learning in urology: a review of the literature on urolithiasis, renal cell carcinoma, and bladder and prostate cancer. World J Urol. 2020 Oct;38(10):2329-2347. doi: 10.1007/s00345-019-03000-5. Epub 2019 Nov 5. PMID 31691082